CLINICAL TRIAL: NCT03243084
Title: Effect of Transcranial Alternating Current Stimulation in Chronic Low Back Pain: A Pilot Study
Brief Title: Transcranial Alternating Current Stimulation in Back Pain- Pilot Sudy
Acronym: BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-0870; R01MH101547 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-01

CONDITIONS: Chronic Low Back Pain
Keywords: tACS; transcranial alternating current stimulation; low back pain; chronic pain; alpha oscillations; heart rate variability
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Each participant will receive sham stimulation and 10Hz tACS stimulation at two separate sessions. The order will be randomized (ie, half the participants will receive sham stimulation at the first session and 10Hz tACS stimulation at the second session, and the other half will receive 10Hz tACS stimulation at the first session and sham stimulation at the second session).
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, meaning that neither the participant nor the experimenter knows what kind of stimulation the participant is receiving. An unblinded monitor (separate from the staff that interacts with the participant) is responsible for creating the stimulation codes that run each session and for ensuring that these codes worked correctly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham tACS (Sham Comparator): Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham.
  Interventions: Device: XCSITE100 Stimulator Sham
- Active 10 Hz tACS (Active Comparator): Participants will receive 2mA of alternating current stimulation at a frequency of 10Hz for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  Interventions: Device: XCSITE100 Stimulator tACS

INTERVENTIONS:
Device: XCSITE100 Stimulator Sham — The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session
  Other Names: Sham tACS
  Arms: Sham tACS
Device: XCSITE100 Stimulator tACS — Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied
  Other Names: tACS
  Arms: Active 10 Hz tACS

SUMMARY:
Chronic pain is a severe disabling problem within society, affecting 25-30% of the United States population.. Transcranial alternating current stimulation (tACS) has the potential to provide a treatment option that is safe, scientifically-supported, low-cost, and easy-to-administer method to effectively reduce symptoms in patients suffering from chronic pain. The purpose of this study is to test the feasibility of using tACS to treat patients with chronic pain, and to collect pilot efficacy as well as EEG and EKG biomarker data for optimizing the design of subsequent large-scale studies. The treatment rationale is to renormalize the presumed pathological structure of alpha oscillations in the prefrontal cortex (PFC) of patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65
* Diagnosed with nonspecific chronic low back pain by clinician
* BMI is less than 30
* Suffered from chronic pain for > 6 months
* Self-report pain measures >4
* Meets criteria for low depression and suicide risk as defined by the Hamilton-Depression Rating Scale
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Not currently taking opioids, benzodiazepines, and anticonvulsant medications

Exclusion Criteria:

* Radicular Pain
* Traumatic brain injury, Any brain devices/implants, including cochlear implants and aneurysm clips
* History of major neurological or psychiatric illness, including epilepsy
* (For females) Pregnancy or breast feeding
* Diagnosis of eating disorder (current or within the past 6 months), Obsessive Compulsive Disorder (lifetime), or Attention-Deficit Hyperactivity Disorder (currently under treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen McCulloch, PhD, DPT, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Plan

REFERENCES:
- [Derived] Prim JH, Ahn S, Davila MI, Alexander ML, McCulloch KL, Frohlich F. Targeting the Autonomic Nervous System Balance in Patients with Chronic Low Back Pain Using Transcranial Alternating Current Stimulation: A Randomized, Crossover, Double-Blind, Placebo-Controlled Pilot Study. J Pain Res. 2019 Dec 11;12:3265-3277. doi: 10.2147/JPR.S208030. eCollection 2019. PMID 31849514
- [Derived] Ahn S, Prim JH, Alexander ML, McCulloch KL, Frohlich F. Identifying and Engaging Neuronal Oscillations by Transcranial Alternating Current Stimulation in Patients With Chronic Low Back Pain: A Randomized, Crossover, Double-Blind, Sham-Controlled Pilot Study. J Pain. 2019 Mar;20(3):277.e1-277.e11. doi: 10.1016/j.jpain.2018.09.004. Epub 2018 Sep 27. PMID 30268803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ran from August 2017 - December 2017. This clinical trial utilized multiple recruitment strategies including UNC University Physical Therapy and Pain clinic locations, informational notify.unc.edu system, and jointheconquest.org along with the listing on clinicaltrials.gov
Groups:
- Sham Then Active 10 Hz tACS: At session 1 this group received sham tACS and at session 2 they received active 10Hz tACS
- Active 10 Hz Then Sham tACS: At session 1 this group received active 10Hz tACS and at session 2 they received sham tACS
Period: Session 1
Arm/Group | Sham Then Active 10 Hz tACS | Active 10 Hz Then Sham tACS
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Washout (1-3 Weeks)
Arm/Group | Sham Then Active 10 Hz tACS | Active 10 Hz Then Sham tACS
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Session 2
Arm/Group | Sham Then Active 10 Hz tACS | Active 10 Hz Then Sham tACS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active 10 Hz Then Sham tACS: At session 1 this group received active 10Hz tACS and at session 2 they received sham 10Hz tACS
- Total: Total of all reporting groups
Arm/Group | Sham Then Active 10 Hz tACS | Active 10 Hz Then Sham tACS | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.8) | 43.4 (13.6) | 43 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.98 (4.1) | 25.92 (5.1) | 25.94 (4.5)
Duration of Pain [Mean (Standard Deviation); unit: years] | 4.8 (3.0) | 9.3 (7.4) | 7.1 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability Before and After 40-minute Stimulation
Description: Changes in parasympathetic tone, increase in high frequency band input via spectral analysis on EKG recordings between active and sham stimulation
Time Frame: before and after 40-minute stimulation at each session
Measure: Mean (Standard Deviation); unit: ms^2
Groups:
- Active10 Hz tACS: Participants will receive 2mA of alternating current stimulation at a frequency of 10Hz for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied
Arm/Group | Sham tACS | Active10 Hz tACS
Number analyzed (Participants) | 20 | 20
ms^2 | 0.206 (0.76) | -0.01 (0.56)
Statistical Analysis 1: Comparison: Sham tACS vs Active10 Hz tACS; A 2x2 ANOVA was used to measure change in HF-HRV by condition (10 Hz vs sham) and session (first vs second) as within subjects variables; Test type: Superiority; p = .319, ANOVA — Threshold for significance is <.05

2. Primary Outcome: Change in Electroencephalogram Power in Alpha Band Before and After 40-minute Stimulation
Description: Changes in the EEG power in the alpha (8-12 Hz) band before and after 40-minute stimulation
Time Frame: 5 minute recordings before and after each 40-minute stimulation at each session.
Measure: Mean (Standard Deviation); unit: square microvolts
Arm/Group | Sham tACS | Active 10 Hz tACS
Number analyzed (Participants) | 20 | 20
square microvolts | 0.03 (0.16) | 0.4 (0.15)

3. Secondary Outcome: Change in Pain Rating on the Visual Analog Scale Before and After 40-minute Stimulation
Description: Self reported pain rating using a Visual Analog Scale (VAS) ranging from 0-10 done before and after stimulation with '0' being no pain and '10' as bad as it could be. Lower values represent a better outcome. (Pain difference was normalized using modulation index to account for ordinal scale)
Time Frame: before and after 40 minute stimulation session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tACS | Active 10 Hz tACS
Number analyzed (Participants) | 20 | 20
units on a scale | -0.178 (0.97) | 0.18 (0.31)
Statistical Analysis 1: Comparison: Sham tACS vs Active 10 Hz tACS; Investigators hypothesized that active stimulation would have a greater normalized pain change using a modulation index [(Pre-Post)/(Pre+Post)]; Test type: Superiority; p = .0488, Wilcoxon (Mann-Whitney) — Threshold for significance is <.05

ADVERSE EVENTS:
Time Frame: Study enrollment until 2 day followup after last session
Description: A side effects questionnaire
Arm/Group | Sham tACS | Active 10 Hz tACS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
Limitations of the study include small sample size. Participants received only 1 session of Active 10 Hz tACS by design but there is likely an additive effect and future studies should investigate multiple sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT03243084/Prot_SAP_000.pdf